CLINICAL TRIAL: NCT00899145
Title: Genetic Modifiers of BRCA1/BRCA2-Related Breast Cancer Risk in BRCA1/BRCA2 Mutation Carriers
Brief Title: Breast Cancer Risk in Women Who Are BRCA1/BRCA2 Mutation Carriers
Status: Withdrawn | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0246; NCI-2009-00608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000590275; GOG-0246 (Other: Gynecologic Oncology Group); GOG-0246 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

GROUPS / COHORTS (1):
- Ancillary-Correlative (biomarker sampling and analysis): Previously collected DNA samples and associated clinical information obtained from BRCA mutation-positive participants enrolled on GOG-0199 are studied. DNA samples are analyzed by mutation testing for variants (i.e., SNPs) in candidate genes of interest. Once genetic testing for a given set of variants has been completed, the coded laboratory data file is merged with selected demographic, clinical, and epidemiological data obtained from the GOG-0199 baseline questionnaire and submitted to the CIMBA Central Database to analyze and publish the data. The epidemiological and SNP data contributed to the central database are then distributed to the investigators responsible for analysis of a particular SNP or set of SNPs from a candidate gene or genetic pathway.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research study is looking at breast cancer risk in women who are BRCA1/BRCA2 mutation carriers. Studying samples of DNA in the laboratory from women who are BRCA1/BRCA2 mutation carriers may help doctors identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVE:

I. To identify potential genetic modifiers of breast cancer risk in women who are carriers of the breast cancer susceptibility genes, BRCA1/2, by collecting data and genetic information from GOG-0199 and contributing it to the Consortium of Investigators of Modifiers of BRCA-Associated Breast Cancer (CIMBA), an international consortium of clinical cancer genetics investigators.

OUTLINE: This is a multicenter study. Patients are stratified by study, country of residence, ethnicity, and birth cohort. Joint analyses of BRCA1 and BRCA2 mutation carriers are further stratified by mutation.

Previously collected DNA samples and associated clinical information obtained from BRCA mutation-positive participants enrolled on GOG-0199 are studied. DNA samples are analyzed by mutation testing for variants (i.e., single nucleotide polymorphisms [SNPs]) in candidate genes of interest. Once genetic testing for a given set of variants has been completed, the coded laboratory data file is merged with selected demographic, clinical, and epidemiological data obtained from the GOG-0199 baseline questionnaire and submitted to the Consortium of Investigators of Modifiers of BRCA-Associated Breast Cancer (CIMBA) Central Database to analyze and publish the data. The epidemiological and SNP data contributed to the central database are then distributed to the investigators responsible for analysis of a particular SNP or set of SNPs from a candidate gene or genetic pathway.

ELIGIBILITY:
Inclusion Criteria:

* Women with or without a personal history of breast cancer prior to enrollment in Gynecologic Oncology Group (GOG)-0199

  * Known currently to be BRCA1/2 mutation carrier either by confirmed outside report or by research testing

    * No BRCA1/2 mutation-negative or mutation-unknown status
* Enrolled on clinical trial GOG-0199 AND meets the following criteria:

  * Completed baseline questionnaire (BQ-199)
  * Provided information on previous breast cancer history, including date of diagnosis
  * Provided complete data from the DNA analysis on the genetic variants of interest
* Available DNA samples for analysis
* Hormone receptor status not specified
* Pre- or post-menopausal status

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Identification of potential genetic modifiers of breast cancer risk | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greene, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States